CLINICAL TRIAL: NCT05335798
Title: Reinforcing CP Robotic Training With Auditory Feedback
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: State University of New York at Buffalo (Other)
Responsible Party: Principal Investigator, Jiyeon Kang, Assistant Professor, State University of New York at Buffalo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00005147
Record Dates: First submitted 2022-03-11; First posted 2022-04-19 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adults with Cerebral Palsy (Experimental): Adults with Cerebral Palsy who are able to be self-ambulatory for minimum 100 feet
  Interventions: Device: Bodyweight augment system; Device: Smart insole

INTERVENTIONS:
Device: Bodyweight augment system — Motorized cables will be providing downward force on the participant's pelvis
Device: Smart insole — Insole provided auditory feedback when heel strike or toe-off events happen

SUMMARY:
The purpose of this study is to create a platform to prolong the adaption obtained from the cable-actuated gait training and encourage the individuals with CP to provide self-care at home.

DETAILED DESCRIPTION:
The experiment protocol involves a maximum of ten sessions and will take two or three hours for each session. Baseline data will be collected before the first session for both overground and treadmill walking. During this session, the sound level will be adjusted based on the feedback received from the users. The researcher will ask the comfortable sound level to the participant before starting the experiment. Training will be conducted on the treadmill with the cable-actuated device for about 20 minutes. When the cables were removed, participants walked on the treadmill for 4 minutes during the post-training session. During training and post-training, participants will be exposed to feedback while walking on the treadmill. After treadmill walking, CP participants will be asked to take a ten-minute break and then practice overground walking for two minutes with auditory feedback (type A) and without it (type B). Effects of 3 different types of auditory feedback will be explored namely, rhythmic sounds, movement sonification, and sound notifying erroneous gait. Group A participants will be further divided into groups depending on the type of auditory feedback that will be provided. Participants will participate in a maximum of 10 sessions, two or three times a week. Before the first and after the last training, participants will be evaluated for functional gait assessment, 6-min-walk, leg strength using a dynamometer, and Modified Ashworth test by a physical therapist.

ELIGIBILITY:
Inclusion Criteria:

* Adults with cerebral palsy (18-65 years old)
* Ambulation of a distance of 100 feet with or without the use of assistive devices.

Exclusion Criteria:

* Severe Equinovarus foot or Genu recurvatum of the knee
* Surgery within 6 months will be excluded.
* Individuals with pregnancy
* Lower limb prosthetics
* Severe respiratory problems such as chronic obstructive pulmonary disease, heart disease, a loss of sensation, uncontrolled blood pressure,
* Seizure disorder
* Severe arthritis

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2021-12-07 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Change of 10m walk between pre/post evaluation and 6 Training sessions | through study completion, an average of 5 weeks
  Timing in seconds during 10 m over ground walking. Lower score means faster (better) walking speed
Change of 6 min walk between Pre/post evaluation | through study completion, an average of 5 weeks
  Measure distance in meter over 6 min walk. Increased distance shows better walking endurance
Change of Ground reaction force between 6 Training sessions | through study completion, an average of 5 weeks
  Bertec Force instrumented treadmill will use to measure vertical ground reaction force in Newton. We will identify whether we can see a distict heel strike and strong push
Change of Kinematics between Pre/post evaluation and 6 Training sessions | through study completion, an average of 5 weeks
  Motion capture data. We will measure hip, knee, and ankle joint angles in degrees. We expect to see If the knees is more extended and dorsiflexion is observed at heel strike the gait is improved
Change of surface electromyography between Pre/post evaluation and 6 Training sessions | through study completion, an average of 5 weeks
  Surface electromyography will be measured for the lower limb. Unit is in mV. We are expecting to measure the peak semg during each gait cycle.

OTHER OUTCOMES:
Change of Muscle tone between Pre/post evaluation | through study completion, an average of 5 weeks
  Modified Ashworth Scale a clinical measure of muscle spasticity. Rated from 0(no increase in muscle tone) to 4(affected part rigid in flexion or extension). Lower score means better muscle tone.
Usability questionnaire of Post evaluation | through study completion, an average of 5 weeks
  Questionnaires were made to understand the the perceived improvement (increased steps and walking speed ) or dose of the intervention (more session and frequency of the intervention). It is rated from 1 very likely to 5 unlikely.
Exit interview after completion of the sessions of Post evaluation | through study completion, an average of 5 weeks
  This is designed for any improvement of future study design. We will ask questions on potential improvement of the intervention
Change of strength of Post evaluation between Pre/post evaluation | through study completion, an average of 5 weeks
  Measure the strength with Dynamometer in N. Higher number means stronger limb.
Change of functional gait assessment between Pre/post evaluation | through study completion, an average of 5 weeks
  Measure different aspects of gait. It is rated from 0 to 3. Higher score means improved improved walking during gait with level surface, change in speed, gait with head turns, step over obstacle, gait with eyes closed, steps.

CONTACTS AND LOCATIONS:
Overall Officials: Jiyeon Kang, Principal Investigator — University at Buffalo
Locations (1):
- University at Buffalo, South Campus, Kimball 115, Buffalo, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified data will be shared upon request to PI.
Time Frame: After the study is completed
Access Criteria: The personnel who is requesting the data needs to explain how the data will be used in their research.

REFERENCES:
- [Background] Chen D, Asaeikheybari G, Chen H, Xu W, Huang MC. Ubiquitous Fall Hazard Identification With Smart Insole. IEEE J Biomed Health Inform. 2021 Jul;25(7):2768-2776. doi: 10.1109/JBHI.2020.3046701. Epub 2021 Jul 27. PMID 33351772
- [Result] Kang J, Martelli D, Vashista V, Martinez-Hernandez I, Kim H, Agrawal SK. Robot-driven downward pelvic pull to improve crouch gait in children with cerebral palsy. Sci Robot. 2017 Jul 26;2(8):eaan2634. doi: 10.1126/scirobotics.aan2634. Epub 2017 Jul 26. PMID 33157884

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT05335798/Prot_SAP_000.pdf
  • Informed Consent Form (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/98/NCT05335798/ICF_001.pdf